CLINICAL TRIAL: NCT01148316
Title: Adaptive Treatment Strategies for Children and Adolescents With Psychiatric Disorders in the Context of Public Health: "Medicine in Practice"
Brief Title: Developing Adaptive Treatment Strategies for Children and Adolescents With Obsessive-compulsive Disorder.
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roseli Shavitt (Other)
Collaborators: University of Pernambuco (Other)
Responsible Party: Sponsor-Investigator, Roseli Shavitt, MD, PhD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPq-HCFMUSP - 259
Record Dates: First submitted 2010-06-02; First posted 2010-06-22 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Developmental Psychiatry; Sequential Randomized Clinical Trial; Obsessive-Compulsive Disorder D009771
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoxetine (Active Comparator): drops or capsules, 10 to 80mg/Day for 14 weeks (first treatment) and as add-on to group CBT non-responders for additional 14 weeks
  Interventions: Drug: fluoxetine
- Group cognitive-behavioral therapy (Active Comparator): weekly, 2 hour sessions with one therapist and one co-therapist for 14 weeks and as add-on to fluoxetine non-responders for additional 14 weeks
  Interventions: Behavioral: Group cognitive-behavioral therapy

INTERVENTIONS:
Drug: fluoxetine — drops or capsules, 10 to 80mg/Day for 14 weeks (first treatment) and as add-on to group CBT non-responders for additional 14 weeks
  Arms: Fluoxetine
Behavioral: Group cognitive-behavioral therapy — weekly, 2 hour sessions with one therapist and one co-therapist for 14 weeks and as add-on to fluoxetine non-responders for additional 14 weeks
  Arms: Group cognitive-behavioral therapy

SUMMARY:
Obsessive-compulsive disorder affects approximately 2% of the population, frequently has its onset during childhood or adolescence and is potentially incapacitating. If not properly treated, this disorder tends to follow a chronic course. Pharmacotherapy with clomipramine and selective serotonin reuptake inhibitors (SSRIs), such as fluvoxamine, fluoxetine and sertraline, has been approved for pediatric OCD. However, up to 30% of patients may not benefit from these treatments, and the presence of residual symptoms is frequent among treatment responders. Cognitive-behavioral therapy (CBT) is also recognized as first line treatment for pediatric OCD, either administered in individual or group format. There is evidence suggesting equivalent efficacy for SSRIs and CBT in pediatric OCD, but there is no data on adaptive treatment strategies regarding such treatments on the long term outcome of OCD patients. The aim of this study is to verify, in a randomized design, if there is an optimal sequential treatment strategy for pediatric OCD, adopting the two most studied treatments for this disorder: an SSRI and group CBT (GCBT). The investigators hypotheses are: (1) both types of treatment will present similar efficacy in the short term (14 weeks); (2) for non-responders to the first type of treatment (fluoxetine up to 80mg/day or GCBT for 14 weeks), combined treatment (fluoxetine + GCBT for another 14 weeks) will be more effective than switching treatment modality (from fluoxetine to GCBT or from GCBT to fluoxetine for additional 14 weeks) after additional 14 weeks.

DETAILED DESCRIPTION:
This is a 28-week open protocol, composed of two phases of randomized treatments with 14 weeks duration.

Inclusion criteria: DSM-IV diagnosis of OCD; age between 7 and 17 years; willing to participate in the protocol; parents or legal tutors agreement with their child participation in the protocol; absence of physical or cognitive impairment that prevent the participation in the protocol.

We expect to end the protocol with 50 patients in each arm (total = 200). For this reason, the purpose is to recruit at least 400 patients for the first randomization (R1: fluoxetine X group CBT). Responders to the initial type of treatment will be maintained in the same procedure for additional 14 weeks. The second randomization (R2) will address non-responders to fluoxetine, who will be randomized to switch to group CBT or receive group CBT as add-on therapy; and non-responders to group CBT, who will be randomized to switch to fluoxetine or receive fluoxetine as add-on therapy.

Fluoxetine will be administered in drops or capsules, in doses ranging from 10 to 80mg/day. Group CBT will be delivered weekly, in 2-hour sessions, in groups of 6 to 8 participants.

At the end of each treatment (weeks 14 and 28), treatment response will be assessed by blind raters, through the YBOCS and CGI-global improvement subscale. Response will be defined as at least 35% reduction in baseline YBOCS scores and a CGI score of 1 or 2.

Efficacy of treatments at the end of R1 will be compared and the efficacy of the different sequences of treatments at the end of R2 (adaptive treatment strategies) will be compared by means of an intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of obsessive-compulsive disorder according to DSM-IV as major problem
* 7 to 17 years
* who agree to participate in the research
* who have parental permission or legal guardian to participate in the research
* that do not have physical or cognitive impairments that prevent the participation of research
* YBOCS ≥ 16 for obsession and compulsion or ≥ 10 for only obsession or compulsion only
* Be above the tenth percentile of weight corresponding to age
* IQ greater than 80 - assessed using the Raven (the screening, if necessary)

Exclusion Criteria:

* Inability to study evaluated adherence to the beginning.
* ANY medical or neurological condition that determines contraindication to any of the treatments or that may influence the evaluation protocol
* pregnancy (women of childbearing age should use contraception)
* Suicidal ideation (with intent) CURRENT

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2010-08; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Treatment response status at week 28 | Yale-Brown Obsessive-Compulsive Scale scores at week 28
  The primary outcome will be the treatment response status, as measured by the variation of Yale-Brown Obsessive-Compulsive Scale,after having received,in a randomized design, different sequential treatments for obsessive-compulsive disorder.
Treatment response status at week 14 | Yale-Brown Obsessive Compulsive Scale Score at week 14
  Treatment resposnse to the first treatment assigned, fluoxetine or group cognitive-behavioral therapy, will be assessed at week 14. Non- responders will be randomized to the second treatment: either combination therapy (fluoxetine plus group cognitive-behavioral therapy) or switch to the other first line treatment (non-responders to fluoxetine as the first treatment switch to group cognitive behavioral therapy and non-responders to cognitive behavioral therapy switch to fluoxetine)

SECONDARY OUTCOMES:
Predictors of treatment response at week 28 | KID-SADS, Family Accomodation Scale, Dimensional Yael-Brown Obsessive-Compulsive Scale
  Socio-demographical and clinical factors, such as gender, age at onset of the disorder, duration of illness, obsessive-compulsive symptom dimensions, psychiatric comorbidities and family accomodation, will be analyzed in relation to the response to the distinct sequential treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Euripedes Miguel, MD, PhD, Principal Investigator — University of Sao Paulo; Roseli G Shavitt, MD, PhD, Study Director — University of Sao Paulo; Guilherme V Polanczyk, MD, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Institue of Psychiatry - Hospital of Clinics - University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Vattimo EFQ, Barros VB, Requena G, Sato JR, Fatori D, Miguel EC, Shavitt RG, Hoexter MQ, Batistuzzo MC. Caudate volume differences among treatment responders, non-responders and controls in children with obsessive-compulsive disorder. Eur Child Adolesc Psychiatry. 2019 Dec;28(12):1607-1617. doi: 10.1007/s00787-019-01320-w. Epub 2019 Apr 10. PMID 30972581